CLINICAL TRIAL: NCT02102711
Title: Oral Vitamin A Supplementation in Neonates With Birth Weight < 1500 g Efficacy and Tolerability in the Prevention of Bronchopulmonary Dysplasia (BDP) and Retinopathy of the Prematurity (ROP)
Brief Title: Oral Vitamin A Supplementation in Neonates With Birth Weight < 1500 g
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesca Garofoli (Other)
Responsible Party: Sponsor-Investigator, Francesca Garofoli, doctor, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITA-1-OS
Record Dates: First submitted 2014-03-06; First posted 2014-04-03 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Bronchopulmonary Dysplasia; Retinopathy of Prematurity
Keywords: VITAMIN A; BLOOD CONCENTRATION; retinopathy of prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Retinopathy of Prematurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitaminA drops (Experimental): 3000 IU/kg/die of Vitamin A oral drops, for 4 weeks.
  Interventions: Dietary Supplement: Vitamin A oral drops
- control (No Intervention): Control of matched infants not supplemented with vitamin A ( beyond standard/routine needed)

INTERVENTIONS:
Dietary Supplement: Vitamin A oral drops
  Other Names: VISPO, BIOTRADING Pharma
  Arms: vitaminA drops

SUMMARY:
Vitamin A is essential for optimal growth, and development. In the newborn, especially if preterm, it is necessary for the cellular differentiation, for the health of the anterior eye, it is a constituent of visual pigment, and it is essential for surfactant synthesis. Immune response Vitamin A supplementation demonstrated to reduces infancy mortality, but very low (<1500g birth weight) and extremely low (<1000g birth weight) preterm infants are born with low body stores of vitamin A and are at high risk of vitamin A deficiency. Nevertheless, optimal vitamin A supplementation for these infants is not clearly defined, despite evidence of benefit of an early supplementation.

Prematurity is associate to the risk for bronchopulmonary dysplasia (BPD) which is a disease marked by respiratory compromise associated with high mortality and severe long-term morbidity, as well as prematurity is associate to the risk for retinopathy, a pathology that may be related to less rhodopsin quantity which seem dependent on vitamin A concentration. Vitamin A can be given enterally, intramuscularly, or intravenously. Recently an oral administration as drops is available resulting particularly convenient avoiding the pain associated with repetitive intramuscular injections, or the discomfort of parenteral administration. Studies of vitamin A in the infant population suggest that plasma retinol concentrations >0.7 µM/L indicate vitamin A sufficiency, nevertheless preterm infants have lower concentration and concentration < 0.35 µM/L are very dangerous. Vitamin A deficiency at this level may constitute a problem for preterm newborn, resulting for example, in histological alterations in the respiratory epithelium leading to chronic lung disease, retinopathy of prematurity, patency of the ductus arteriosis, and immune competence deficiency.

The aim of the present study is to verify efficacy and tolerability of a new oral administration of vitamin A as drops, 3000 IU/kg/die for 4 weeks, in infants < 1500g weight at birth, verifying the competence of the supplementation reaching ideal blood concentration (≥0.7 µM/L) and relating the blood achieved concentrations of vitamin A to the outcome in typical pathologies, as BPD and ROP. Not treated group of matched newborn infants is the controlarm.

ELIGIBILITY:
Inclusion Criteria:

* parents signed informed consent
* very low birth weight infants undergoing ventilation for at least 24 hours
* Infants able to receive adequate breast or formula milk

Exclusion Criteria:

* parents denied informed consent
* congenital malformations
* infants not able to receive breast or formula milk

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Vitamin A blood concentration (µM/L) | participants will be followed for the duration of Vitamin A oral administration, an expected average of 4 weeks
  Vitamin A functional concentration

SECONDARY OUTCOMES:
number of bronchopulmonary dysplasia and of retinopathy of prematurity | 1 year
  number of events

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Stronati, MD, Study Director — IRCCS Policlinico S. Matteo, Pavia, Italy
Locations (2):
- Italy (2):
  - IRCCS Policlinico S. Matteo, Pavia, PV
  - IRCCS Policlinico S.Matteo; Neonatal Intensive Care Unit, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garofoli F, Barilla D, Angelini M, Mazzucchelli I, De Silvestri A, Guagliano R, Decembrino L, Tzialla C. Oral vitamin A supplementation for ROP prevention in VLBW preterm infants. Ital J Pediatr. 2020 Jun 3;46(1):77. doi: 10.1186/s13052-020-00837-0. PMID 32493448